CLINICAL TRIAL: NCT03905876
Title: Psychological Experience of the End of the Treatment During a Clincal Trial of the Early Phase and Role of the Initial prédispositions ( VRAIMENT)
Brief Title: Psychological Experience of Discontinuation an Early Phase Treatment by Patients
Acronym: VRAIMENT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut du Cancer de Montpellier - Val d'Aurelle (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2018-A02330-55
Record Dates: First submitted 2019-01-29; First posted 2019-04-05 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2024-10

CONDITIONS: Psychological Distress; Cancer
Keywords: Psychological experience; early clinical trial; initial predisposition
MeSH Terms: conditions — Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- assessment of psychological experience (Other): Questionnaire
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Questionnaire to evaluate psychological experience

SUMMARY:
While there is currently some study on the motivations and experiences of patients integrating early phase clinical trials, to our knowledge, no study has explored the future of patients coming out of these trials. It is therefore urgent to better understand the feelings and experiences of patients who discontinue their treatment in a clinical trial of early phase (EP) to provide them with tailored and personalized support. In addition, the end of treatment may have a different impact on the person depending on whether the treatment was discontinued due to the protocol (the patient received the full treatment as planned) or to an early withdrawal (intolerable toxicities or progression of the disease).

DETAILED DESCRIPTION:
EP trials are crucial in the development of a new cancer treatment. Given the side effects and limited knowledge of any new treatment, the inclusion of patients in this EP faces ethical barriers and communication barriers. This is all the more true as EPs are generally aimed at patients with advanced cancer. Also, faced with these different issues, volunteer patients usually have ambivalent motives. Catt and his collaborators have shown that the primary motivations for agreeing to integrate an early phase are the medical benefits, then the best option available, the maintenance of hope and only then, the aid to research.

And more, at the beginning of a EP trial, most patients simultaneously experience multiple complex symptoms related to their cancer or treatment. These symptoms and their functional consequences generate psychological distress and reduce their quality of life related to health. Measuring psychological distress and quality of life before entering a clinical trial is therefore essential for the analysis of psychopathological processes.

Since emotional regulation involves many aspects, it seems scientifically relevant to choose central scales, which cover broad psychopathological functions, to capture the psychological distress of patients. This battery of scales should include an assessment of levels of anxiety, depression and anger (as markers of irritability) but also pre-morbid psychological predispositions. Indeed, some variables such as resilience and optimism are known to influence the level of psychopathological symptomatology and the experience of cancer. Finally, qualitative interviews would better capture the experience of patients with advanced cancer when they are confronted with an end of treatment in EP.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven solid cancer locally advanced or metastatic in treatment failure with standard treatments
* Antitumor therapy in an early phase clinical trial
* Comprehension in French sufficient for a good completion of the questionnaires
* Informed consent signed before any specific procedure to study
* Belong to a French social security scheme or equivalent scheme
* Age ≥ 18 years

Exclusion Criteria:

* Score <15 on the Montreal Cognitive Assessment (MoCA) test assessing overall cognitive functioning
* Presence of proven psychiatric disorders (eg, mental retardation, psychotic disorders, learning disabilities, attention deficit / hyperactivity disorder, bipolar disorder ...), excluding reactional mood disorders to the experience of the disease, or receiving treatment psychotropic disorder that ability of reasoning, judgment or understanding
* Possibility of benefiting from standard therapeutic options
* Included in an exclusive clinical trial or for which the sponsor has refused to that his trial are associate to the study "VRAIMENT"
* Physical inability to answer questionnaires
* Legal incapacity or limited legal capacity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2019-01-21 (Actual); Primary Completion 2024-04-04 (Actual); Study Completion 2024-04-04 (Actual)

PRIMARY OUTCOMES:
Score of anxiety and depression at the end of treatement in an early clinical phase by using the scale HADS (hospital anxiety and depression scale). The range is 0 to 21. The severe anxiety or depression is 21. | Approximatey 36 months
  Comparison of the questionnaires collected at the time of inclusion and end of treatment in an early clinical phase

SECONDARY OUTCOMES:
Anxiety score obtained by using the HADS subscale (hospital anxiety and depression scale). The range is 0 to 21. | Day 1 and approximately 36 months
  Baseline and end of treatment
Depression score obtained by using the HADS subscale (hospital anxiety and depression scale). The range is 0 to 21. | Day 1 and approximately 36 months
  Baseline and end of treatment
Anger assessed by using the STAXI-2 questionnaire (stait-trait anger expression inventory) | Day 1 and approximately 36 months
  Baseline and end of treatment
Optimism assessed by using the optimism scale (the Life Orientation Test-Revised - LOT-R) . The range is 0 to 40. | Day 1
  Baseline
Resilience assessed by using the resilience score (the Connor-Davidson Resilience Scale - CD-RICS-10). The range is 0 to 40. | Day 1
  Baseline
Overall quality of life score assessed by the EORTC (european organization for research and treatment of cancer) questionnaire QLQ-C30 (quality questionnaire) | Day 1 and approximately 36 months
  Baseline and end of treatment
Reason for discontinuation of trial (i.e., intolerable toxicity, disease progression or termination of the protocol as described in the trial) | approximately 36 months
  End of treament
Language markers through 3 main contents: 1/ the experience of the study exit, 2/ the representations of the clinical trial in which the patient participated and 3/ his future. | Day 1 and approximately 36 months
  Baseline and end of treatment
Motivation assessed by using a motivation questionnaire | Day 1
  Baseline

CONTACTS AND LOCATIONS:
Overall Officials: jean Pierre BLEUSE, Dr, Study Director — Insititut régional de Cancer de Montpellier
Locations (1):
- Institut régional du Cancer de Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jenkins V, Solis-Trapala I, Langridge C, Catt S, Talbot DC, Fallowfield LJ. What oncologists believe they said and what patients believe they heard: an analysis of phase I trial discussions. J Clin Oncol. 2011 Jan 1;29(1):61-8. doi: 10.1200/JCO.2010.30.0814. Epub 2010 Nov 22. PMID 21098322
- [Background] Bredart A, Bodson S, Le Tourneau C, Flahault C, Bonnetain F, Beaudeau A, Coquan E, Dolbeault S, Paoletti X. Patients' perceived tolerance of side effects in phase I cancer clinical trials: A qualitative study. Eur J Cancer Care (Engl). 2017 Nov;26(6). doi: 10.1111/ecc.12596. Epub 2016 Oct 12. PMID 27734561
- [Background] Kroenke K, Johns SA, Theobald D, Wu J, Tu W. Somatic symptoms in cancer patients trajectory over 12 months and impact on functional status and disability. Support Care Cancer. 2013 Mar;21(3):765-73. doi: 10.1007/s00520-012-1578-5. Epub 2012 Sep 1. PMID 22941116
- [Background] Catt S, Langridge C, Fallowfield L, Talbot DC, Jenkins V. Reasons given by patients for participating, or not, in Phase 1 cancer trials. Eur J Cancer. 2011 Jul;47(10):1490-7. doi: 10.1016/j.ejca.2011.02.020. Epub 2011 Mar 30. PMID 21454072
- [Background] Balbuena L, Bowen R, Baetz M, Marwaha S. Mood Instability and Irritability as Core Symptoms of Major Depression: An Exploration Using Rasch Analysis. Front Psychiatry. 2016 Oct 26;7:174. doi: 10.3389/fpsyt.2016.00174. eCollection 2016. PMID 27833568
- [Background] Tian J, Hong JS. Assessment of the relationship between resilience and quality of life in patients with digestive cancer. World J Gastroenterol. 2014 Dec 28;20(48):18439-44. doi: 10.3748/wjg.v20.i48.18439. PMID 25561814
- [Background] Matzka M, Mayer H, Kock-Hodi S, Moses-Passini C, Dubey C, Jahn P, Schneeweiss S, Eicher M. Relationship between Resilience, Psychological Distress and Physical Activity in Cancer Patients: A Cross-Sectional Observation Study. PLoS One. 2016 Apr 28;11(4):e0154496. doi: 10.1371/journal.pone.0154496. eCollection 2016. PMID 27124466
- [Background] Bozo O, Gundogdu E, Buyukasik-Colak C. The moderating role of different sources of perceived social support on the dispositional optimism-- posttraumatic growth relationship in postoperative breast cancer patients. J Health Psychol. 2009 Oct;14(7):1009-20. doi: 10.1177/1359105309342295. PMID 19786527